CLINICAL TRIAL: NCT02573857
Title: A Phase Ib Study to Characterise the Antimalarial and Transmission Blocking Activity of a Single Dose of DSM265 or OZ439 in Healthy Subjects With Induced Blood Stage Plasmodium Falciparum or Plasmodium Vivax Infection
Brief Title: A Study to Characterise the Antimalarial and Transmission Blocking Activity of a Single Dose of DSM265 or OZ439 in Healthy Subjects With Induced Blood Stage Plasmodium Falciparum or Plasmodium Vivax Infection
Acronym: DSMOZ-2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry); Q-Pharm Pty Limited (Industry); Queensland Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QP15C11
Record Dates: First submitted 2015-10-06; First posted 2015-10-12 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Malaria
Keywords: Induced blood stage malaria; Transmission; Gametocytemia
MeSH Terms: conditions — Malaria | interventions — DSM265; artefenomel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DSM265 P. falciparum (Experimental): Cohort 1: the efficacy of a single administration of 400 mg DSM265 for the clearance of asexual blood stages of P. falciparum will be determined. Activity of a second single dose of 400 mg DSM265 against gametocytes will be assessed in this cohort only if sexual stages are identified by PCR following the initial drug treatment.
  Interventions: Drug: DSM265
- OZ439 P. vivax (Experimental): Cohort 2: subjects will be infected with P. vivax by IBSM, then treated with a single 200 mg dose OZ439. If recrudescence occurs following initial drug treatment with 200 mg OZ439, then affected participants who reach the treatment threshold will receive a single 400 mg dose of OZ439.
  Interventions: Drug: OZ439
- DSM265 P. vivax (Experimental): Cohort 3: subjects will be infected with P. vivax by IBSM, then treated with a single 400 mg dose of DSM265
  Interventions: Drug: DSM265

INTERVENTIONS:
Drug: DSM265 — Oral suspension from bulk powder
  Arms: DSM265 P. falciparum; DSM265 P. vivax
Drug: OZ439 — Oral suspension from powder in a bottle
  Other Names: Artefenomel
  Arms: OZ439 P. vivax

SUMMARY:
Part A

-Cohort 1 DSM265 will be administered as a single dose (400 mg). For cohort 1 only, an additional single dose (400 mg) of DSM265 may be given if gametocytemia develops. Treatment with DSM265 will be given after an overnight fasting period of ≥ 8 hours. If dosing is to occur in the evening, subjects will be required to fast for ≥4 hours prior to receiving treatment. Subjects will be required to fast for a further four hours anytime after dosing with DSM265.

Part B

* Cohort 2 OZ439 will be administered as a single 200 mg dose. If recrudescence is observed, a single 400 mg dose of OZ439 will be given. Treatment with OZ439 will be administered after an overnight fasting period of ≥ 6 hours. If dosing is to occur in the evening, subjects will be required to fast for ≥4 hours prior to receiving treatment. Participants will drink 200 mL of milk prior to drug administration, and then swallow the appropriate volume of OZ439 suspension. Subjects will be required to fast for a further six hours anytime after dosing with OZ439.
* Cohort 3 DSM265 will be administered as a single dose (400 mg) as described for cohort 1. No additional dose will be administered.

DETAILED DESCRIPTION:
This is a single-centre, open label study using induced blood stage malaria (IBSM) infection to assess the effectiveness of the investigational drugs DSM265 or OZ439 in reducing parasitemia. Transmission blocking activity of DSM265 (in P. falciparum infection; cohort 1 only) and infectivity to vector mosquitoes prior to drug treatment (in P. vivax infection; cohort 2 and 3) will also be assessed. This study will be conducted in up to three cohorts (n = 8 per cohort), and will be divided into 2 parts. In Part A (cohort 1) the efficacy of a single administration of 400 mg DSM265 for the clearance of asexual blood stages of P. falciparum will be determined. Activity of a second single dose of 400 mg DSM265 against gametocytes will be assessed in this cohort only if sexual stages are identified by PCR following the initial drug treatment. In Part B, subjects will be infected with P. vivax by IBSM, then treated with a single 200 mg dose OZ439 (cohort 2) or 400 mg dose of DSM265 (cohort 3). For cohort 2, if recrudescence occurs following initial drug treatment with 200 mg OZ439, then affected participants who reach the treatment threshold will receive a single 400 mg dose of OZ439. The PK/PD relationship following drug treatment will be determined in order to further characterize the antimalarial activity of the investigational drug in the IBSM system using P. falciparum (for cohort 1; 400 mg DSM265) or P. vivax (for cohort 2, 200 mg OZ439; cohort 3, 400 mg DSM265).

The treatment effects on gametocytemia (if sexual blood stages are detected by PCR) and transmission blocking activity of DSM265 will be investigated as a secondary objective for cohort 1 (P. falciparum infection). Prior to drug treatment, the infectivity of P. vivax IBSM infection to vector mosquitoes will also be investigated as a secondary objective for Part B, cohorts 2 and 3. The exposures achieved with the doses proposed for DSM265 used in Part A and DSM265 or OZ439 in Part B are associated with a safety profile which is well described from previous studies and significantly below the maximum tolerated exposures reported for either drug.

ELIGIBILITY:
Inclusion Criteria:

Health status:

* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 5 minutes resting in supine position:

  * 90 mmHg < systolic blood pressure (SBP) <140 mmHg,
  * 50 mmHg < diastolic blood pressure (DBP) <90 mmHg,
  * 40 bpm< heart rate (HR) <100 bpm.
* Normal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position, QTcF≤450 ms (males and females) with absence of second or third degree atrioventricular block or abnormal T wave morphology.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy participants enrolled in this clinical investigation. More specifically for serum creatinine, hepatic transaminase enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the Participant has documented Gilbert syndrome) should not exceed the upper laboratory norm and haemoglobin must be equal or higher than the lower limit of the normal range
* As there is the risk of adverse effects of the investigational drugs (DSM265 and OZ439), and standard curative treatment (Riamet and primaquine - cohort 1 only) in pregnancy, it is important that any participants involved in this study do not get pregnant or get their female partners pregnant (refer to Section 6.7).

For cohort 1 and 3 (treatment with DSM265):

Female participants of childbearing potential (WOCBP) may be enrolled in the DSM265 cohorts but must have adequate contraception in place for the duration of the study and up to 60 days (9 weeks) after the last dose of DSM265, with adequate contraception defined as:

* Stable hormonal contraception (with an approved oral, transdermal or depot regimen) for at least 3 months prior to screening i.e. oral contraceptives, either combined or progestogen alone, hormonal implantable contraception, vaginal ring, contraceptive patches
* Intrauterine (IUD) device or system in place for at least 3 months prior to screening
* Male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant Abstinent female participants must agree to start a double method if they start a sexual relationship during the study and for up to 60 days (9 weeks) following the last dose of DSM265.

Male participants to be dosed with DSM265 in cohort 1 or 3 must agree to use a double method of contraception including condom plus diaphragm or condom plus stable oral/transdermal/injectable hormonal contraceptive by female partner from at least 14 days prior to the time of the dose of the study drug through 120 days (17 weeks) after the last dose of DSM265.

Abstinent male participants must agree to start a double method if they start a sexual relationship during the study and for up to 120 days (17 weeks) weeks following the last dose of DSM265.

For cohort 2 (treatment with OZ439):

Female subjects must be considered as women of not childbearing potential (WONCBP) to be eligible. WONCBP is defined as:

* Spontaneous amenorrhoea for at least 1 year or spontaneous amenorrhea for at least 6 months confirmed by an FSH result above the laboratory defined range for post-menopausal
* or permanently sterilised (eg tubal occlusion, hysterectomy, bilateral salpingectomy) Female subjects with same sex partners (abstinence from penile-vaginal intercourse), are eligible when this is their preferred and usual lifestyle.

Male participants to be dosed with OZ439 in cohort 2 must agree to use a double method of contraception including condom plus diaphragm or condom plus stable oral/transdermal/injectable hormonal contraceptive by female partner from at least 14 days prior to the time of the dose of the study drug through 96 days (14 weeks) after the last dose of OZ439.

Abstinent male participants must agree to start a double method if they start a sexual relationship during the study and for up to 96 days (14 weeks) following the last dose of OZ439.

For Part B only (cohort 2 and 3):

- All subjects must be Duffy Blood group positive. Female subjects of childbearing potential (Cohort 3 only) should be blood group Rh positive.

Regulations:

- Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

Medical history and clinical status:

* Any history of malaria or participation to a previous malaria challenge study
* Must not have travelled to or lived in a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.
* Has evidence of increased cardiovascular disease risk (defined as >10%, 5 year risk) as determined by the Australian Absolute Cardiovascular Disease Risk Calculator (http://www.cvdcheck.org.au/). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, total and HDL cholesterol (mmol/L), and reported diabetes status.
* History of splenectomy.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion.
* Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin-dependent and non-insulin dependent diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive compulsive disorder
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within 5 years of screening, regardless of whether there is evidence of local recurrence or metastases
* Participants with history of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis including depression or receiving psychiatric drugs or who has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Frequent headaches and/or migraine, recurrent nausea, and/or vomiting (more than twice a month)
* Presence of acute infectious disease or fever (e.g., sub-lingual temperature ≥ 38.5°C) within the five days prior to inoculation with malaria parasites.
* Evidence of acute illness within the four weeks before trial prior to screening that the Investigator deems may compromise subject safety.
* Significant inter-current disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
* Participant has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhoea.
* Participation in any investigational product study within the 12 weeks preceding the study.
* Blood donation, any volume, within 1 month before inclusion or participation in any research study involving blood sampling (more than 450 mL/ unit of blood), or blood donation to Red Cross (or other) blood bank during the 8 weeks preceding the reference drug dose in the study.
* Participant unwilling to defer blood donations to the Australian Red Cross Blood Service (ARCBS) for 6 months.
* Medical requirement for intravenous immunoglobulin or blood transfusions.
* Participant who has ever received a blood transfusion.
* Symptomatic postural hypotension at screening, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 minutes when changing from supine to standing position.
* History or presence of alcohol abuse (alcohol consumption more than 40 g per day) or drug habituation, or any prior intravenous usage of an illicit substance.
* Smoking more than 5 cigarettes or equivalent per day and unable to stop smoking for the duration of the study.
* Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (participants will be advised by phone not to consume any poppy seeds in this time period).
* Excessive consumption of beverages containing xanthine bases, including Red Bull, chocolate etc. more than 400 mg caffeine per day (equivalent to more than 4 cups per day)

Interfering substance:

* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life (whichever is longer) of the medication
* Any vaccination within the last 28 days.
* Any corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants. Any participant currently receiving or having previously received immunosuppressive therapy, including systemic steroids including adrenocorticotrophic hormone (ACTH) or inhaled steroids in dosages which are associated with hypothalamic-pituitary-adrenal axis suppression such as 1 mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids (budesonide 800 μg per day or fluticasone 750 μg).
* Any recent (< 6 weeks) or current systemic therapy with an antibiotic or drug with potential anti-malarial activity (i.e. chloroquine, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, hydroxychloroquine, etc.)

General conditions:

* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or is unable to cooperate because of a language or mental deficit.
* Any participant in the exclusion period of a previous study according to applicable regulations.
* Any participant who lives alone (from Day 0 until at least the end of the anti-malarial drug treatment).
* Any participant who cannot be contacted in case of emergency for the duration of the trial and up to 2 weeks following end of study visit.
* Any participant who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Any participant without a good peripheral venous access.

Biological status

* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-hepatitis A or E virus (IgM) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab)
* Any drug listed in Table 2 (Drug Screening) in the urine drug screen unless there is an explanation acceptable to the medical investigator (e.g., the participant has stated in advance that they consumed a prescription or OTC product which contained the detected drug) and/or the Participant has a negative urine drug screen on retest by the pathology laboratory.

Specific to the study_

* Cardiac/QT risk

  * Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
  * History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia. Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia, or hypomagnesaemia.
  * Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analyses on study
* Known hypersensitivity to DSM265 or OZ439, or any of its excipients or 4-aminoquinolines, artemether or other artemisinin derivatives, lumefantrine, or other arylaminoalcohols.
* Known severe reaction to mosquito bites other than local itching and redness.
* Unwillingness to abstain from consumption of citrus (grapefruit, Seville orange, etc.) for ≥21 days prior to initiation of the study (inoculation; Day 0) and for the study duration.
* Unwillingness to abstain from consumption of quinine containing foods/beverages such as tonic water, lemon bitter, from inoculation (Day 0) to the end of the malaria treatment.
* Any history or presence of lactose intolerance.
* Use of prescription drugs, herbal supplements, within four weeks prior to administration of the study drug, and/or over-the-counter (OTC) medication, dietary supplements (including vitamins) within two weeks prior to initial dosing (Note: diazepam interferes with the analysis of blood levels of DSM265 and thus should not have been used for at least 8 weeks prior to administration of the study drug). If needed (i.e. an incidental and limited need) paracetamol is acceptable up to 4 g/day.

Participants are requested to refrain from taking non-approved concomitant medication from recruitment until the conclusion of the study.

Participants who are excluded from participation on study days for any of the above reasons may be eligible to participate on a postponed schedule if the Investigator considers this appropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Prof, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Q-Pharm Clinics, Herston, Queensland, Australia

REFERENCES:
- [Derived] Dini S, Zaloumis SG, Price DJ, Gobeau N, Kummel A, Cherkaoui M, Moehrle JJ, McCarthy JS, Simpson JA. Seeking an optimal dosing regimen for OZ439/DSM265 combination therapy for treating uncomplicated falciparum malaria. J Antimicrob Chemother. 2021 Aug 12;76(9):2325-2334. doi: 10.1093/jac/dkab181. PMID 34179977
- [Derived] Collins KA, Abd-Rahman AN, Marquart L, Ballard E, Gobeau N, Griffin P, Chalon S, Mohrle JJ, McCarthy JS. Antimalarial Activity of Artefenomel Against Asexual Parasites and Transmissible Gametocytes During Experimental Blood-Stage Plasmodium vivax Infection. J Infect Dis. 2022 Mar 15;225(6):1062-1069. doi: 10.1093/infdis/jiaa287. PMID 32479608
- [Derived] Collins KA, Ruckle T, Elliott S, Marquart L, Ballard E, Chalon S, Griffin P, Mohrle JJ, McCarthy JS. DSM265 at 400 Milligrams Clears Asexual Stage Parasites but Not Mature Gametocytes from the Blood of Healthy Subjects Experimentally Infected with Plasmodium falciparum. Antimicrob Agents Chemother. 2019 Mar 27;63(4):e01837-18. doi: 10.1128/AAC.01837-18. Print 2019 Apr. PMID 30858218

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After reviewing the safety data obtained from the first 2 cohorts, the SRT decided not to enrol Cohort 3.
Period: Overall Study
Arm/Group | DSM265 P. Falciparum | OZ439 P. Vivax
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSM265 P. Falciparum | OZ439 P. Vivax | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (4) | 24.9 (4.6) | 24.8 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.4 (2) | 22.6 (2.8) | 23 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (PRR) of DSM265 or OZ439
Description: Efficacy of a single 400 mg dose of DSM265 or a 200mg dose of OZ439. The primary efficacy variable is parasite reduction ratio (PRR) of asexual parasites based on qPCR analysis of blood level parasitemia pre-dose and following administration of study drug.
  The parasite reduction ratio (PRR) provides an estimate of the efficacy of an antimalarial treatment and is the ratio of the parasite density between admission and 48 h post antimalarial treatment.
Time Frame: From baseline to 48 hours post antimalarial treatment
Population: Subject R104 in Cohort 1 was excluded from PRR analysis because parasitaemia was not observed in this subject.
Measure: Mean (95% Confidence Interval); unit: PRR
Arm/Group | DSM265 P. Falciparum | OZ439 P. Vivax
Number analyzed (Participants) | 7 | 8
PRR | 603 [410 to 886] | 46 [36 to 61]

2. Primary Outcome: Efficacy of OZ439 on P. Vivax
Time Frame: From baseline to 48 hours post antimalarial treatment
Population: Redundant outcome measure. Results are reported in Outcome Measure 1 (Efficacy (PRR) of DSM265 or OZ439).
Arm/Group | DSM265 P. Falciparum | OZ439 P. Vivax
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Safety of DSM265 or OZ439 - Number of Adverse Events
Description: Assessement of Adverse Events (AE) (unexpected toxicities, adverse events encountered during or after investigational drug administration)
Time Frame: From challenge inoculum (day 0) up to day 28 (+/-3 days)
Measure: Number; unit: Number of adverse events
Arm/Group | DSM265 P. Falciparum | OZ439 P. Vivax
Number analyzed (Participants) | 8 | 8
Number of adverse events | 53 | 107

4. Secondary Outcome: Gametocytemia Clearance With DSM265
Time Frame: From Drug administration up to day 28 (+/-3 days) following inoculum
Reporting Status: Not Posted

5. Secondary Outcome: P. Vivax Transmission
Time Frame: From challenge inoculum (day 0) and up to day 28 (+/-3 days)
Reporting Status: Not Posted

6. Secondary Outcome: Parasite Density (Parasite/ml) Assessed by qPCR
Time Frame: From From drug administration until Standard of Care administration, or up to day 28 (+/-3 days)
Reporting Status: Not Posted

7. Secondary Outcome: Drug Concentration (PK) (ng/ml)
Time Frame: From From drug administration until Standard of Care administration, or up to day 28 (+/-3 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Until end of study, 28 +/- 3 days
Arm/Group | DSM265 P. Falciparum | OZ439 P. Vivax
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSM265 P. Falciparum (N=8) | OZ439 P. Vivax (N=8)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Administration site haematoma (General disorders) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (4)
Fatigue (General disorders) | 3 (3) | 3 (6)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 3 (4) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 8 (24)
Vessel puncture site thrombosis (General disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (10)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 5 (5)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 4 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (8) | 6 (19)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less